CLINICAL TRIAL: NCT01024725
Title: Evaluation of a Vaccination Campaign With A(H1N1)v Pandemic Vaccines: a Prospective Cohort Study
Brief Title: Evaluation of Pandemic Vaccination Campaign
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Sponsor
Other Study IDs: AH1N1-483-09THL; EudraCT 2009-015700-26 (Other: NAM Finland); ETL R09152M
Record Dates: First submitted 2009-11-02; First posted 2009-12-03 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Influenza Caused by the Novel A(H1N1)v Influenza Virus
Keywords: A(H1N1)v influenza; vaccination; pandemic

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal/oral swabs, serum samples and peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Not (yet) vaccinated persons: The participants do not want to take the vaccine (available only in the national vaccination campaign) or have not received it yet
  Interventions: Other: Follow-up
- Vaccinated persons: The participants have taken the vaccine according to the national vaccination campaign
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Nasopharyngeal/oropharyngeal and blood samples, interviews, questionnaires, register data

SUMMARY:
A cohort of 4000 community-dwelling adults is followed to evaluate the effectiveness of the Finnish national A(H1N1)v influenza vaccination campaign in preventing the first episode of laboratory-confirmed A(H1N1)v influenza. The safety of vaccination and the severity of the disease are followed primarily from health care registers. In a subgroup of 200 participants, the humoral and cellular immunogenicity of the vaccine will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Full legal competence;
* Written informed consent obtained;
* Assigned to use the services of Tampere health centre and community-dwelling;
* At least 18 and no more than 75 years old, inclusive;
* Belongs to the target group of A(H1N1)v vaccination in the region during the pandemic vaccination campaign;
* Able to communicate fluently in Finnish or Swedish
* Able to adhere to all protocol required study procedures without any special burden or risk, as judged by the investigator or designate.

Exclusion Criteria:

* For the total study cohort, no specific exclusion criteria will be applied;
* For the subgroup for follow-up of immunogenicity of the vaccine (immunogenicity cohort), exclusion criteria comprise:

  * previous severe allergic reaction to influenza vaccines or known severe allergy to the ingredients of the vaccine
  * previous severe allergic reaction to eggs
  * significant immunological disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will be invited from the population assigned to use the services of Tampere health centre, according to the target groups for pandemic vaccination. Invitations will be distributed at the maternity clinics for pregnant women, at work places for health professionals, and letters will be sent home to random sample of subjects at age groups of 18-24 years, 25-64 years and potetially later at 65-75 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 3518 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of vaccination in preventing the first episode of laboratory-confirmed A(H1N1)v infection in adults | 3 November 2009 to 30 April 2010

SECONDARY OUTCOMES:
Safety of vaccination with the A(H1N1)v vaccine | 3 November 2009 to 31 October-November 2010
Severity and possible complications of the A(H1N1)v influenza | 3 November 2009 to 31 October-November 2010
Humoral and cellular immune responses to the vaccine (subgroup of 200 adults) | 3 November 2009 to 31 October-November 2010
Effectiveness of the vaccine in subgroups | 3 November 2009 to 31 October-November 2010

CONTACTS AND LOCATIONS:
Overall Officials: Terhi M Kilpi, MD PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Tampere, Finland

REFERENCES:
- [Derived] Syrjanen RK, Jokinen J, Ziegler T, Sundman J, Lahdenkari M, Julkunen I, Kilpi TM. Effectiveness of pandemic and seasonal influenza vaccines in preventing laboratory-confirmed influenza in adults: a clinical cohort study during epidemic seasons 2009-2010 and 2010-2011 in Finland. PLoS One. 2014 Sep 29;9(9):e108538. doi: 10.1371/journal.pone.0108538. eCollection 2014. PMID 25265186